CLINICAL TRIAL: NCT00302705
Title: Prospective, Randomized, Open-Label Study in Patients With Mild-to-Moderate Essential Hypertension to Compare the Antihypertensive Efficacy Determined by Ambulatory Blood Pressure Monitoring of Valsartan and Enalapril After Missing One Dose
Brief Title: Comparison of the Antihypertensive Efficacy of Valsartan and Enalapril After Missing One Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Vigo (Other)
Collaborators: Hospital Clinico Universitario de Santiago (Other); Novartis (Industry)
Responsible Party: Ramon C. Hermida, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAL-489A2425; 2004-001725-25
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Hypertension
Keywords: Ambulatory blood pressure monitoring; Valsartan; Enalapril; Missing dose
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Enalapril; Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valsartan (Active Comparator): 160 mg/day on awakening
  Interventions: Drug: Valsartan, Enalapril; Device: Ambulatory blood pressure monitoring; Procedure: Missing one dose
- Enalapril (Active Comparator): 10-20 mg/day on awakening
  Interventions: Drug: Valsartan, Enalapril; Device: Ambulatory blood pressure monitoring; Procedure: Missing one dose

INTERVENTIONS:
Drug: Valsartan, Enalapril — 160 mg valsartan versus 10-20 mg enalapril
Device: Ambulatory blood pressure monitoring — Blood pressure measured at 20-min intervals from 07:00 to 23:00 hours and at 30-min intervals at night for 48 consecutive hours
Procedure: Missing one dose — Patients skip the dose the second day of monitoring

SUMMARY:
This study was designed in order to evaluate the blood pressure lowering effect of valsartan compared to enalapril over 24 hours after skipping one daily dose. Both drugs act on the renin-angiotensin-aldosterone system (RAAS) and are widely use for the treatment of hypertension. Previous studies had a significant limitation: the effect of a missing dose was not evaluated after the whole 24 hours post missing dose period (48 hours after last taken dose), and as a result, it does not imitate the real life situation of a missing dose.

DETAILED DESCRIPTION:
The incidence of cardiovascular events, such as myocardial infarction, sudden cardiac death, ventricular arrhythmias, stroke, myocardial ischemia and angina pectoris, reaches the peak during the early morning hours. This period corresponds with the sharp increase in heart rate (HR) and blood pressure (BP) (morning BP surge) which takes place upon arising form overnight sleep. Furthermore, the RAAS is activated in the morning, and may contribute to morning BP surge and to morning increase in cardiovascular risk. BP control over the entire 24 hours dosing interval, including the early morning period (18 - 24 hrs post-dosing) is critical in order to prevent cardiovascular events, thus providing a better protection to patients with essential hypertension. Apart from the significance of establishing the 24-hour BP lowering effect of an antihypertensive drug, it is fundamental to further investigate the effect of a missing dose. Approximately 15 to 20% of hypertensive patients do not recall to take their medication in average 3 days every month. During these periods, patients could be on a higher risk of having a cardiovascular event resulting in a poorer long-term prognosis. Therefore, it is crucial to establish the BP lowering effect of the antihypertensive treatment beyond 24-hour of dose intake. Ambulatory blood pressure monitoring (ABPM) has proven advantages compared to conventional BP measurement and ambulatory BP levels are closely associated with target organ damage and clinical cardiovascular events in hypertensive patients. However most of the studies using this technique have been conducted with monitoring for a 24-hour period. In this study 48-hour ABPM will be utilized in order to investigate the antihypertensive effect beyond 24 hours. This study was designed in order to evaluate the BP lowering effect of valsartan compared to enalapril over 24 hours after skipping one daily dose. Both drugs act on the RAAS and are widely use for the treatment of hypertension. Enalapril was selected since a previous similar study was performed using it as a comparison drug. An 8-week study with candesartan and enalapril was done to evaluate their antihypertensive efficacy and their effect duration. However, this study had a significant limitation, the effect of a missing dose was not evaluated after the whole 24 hours post missing dose period (48 hours after last taken dose), and as a result, it does not imitate the real life situation of a missing dose. Therefore, we decided to perform the present study with the purpose of further investigate the effect of these antihypertensive treatments beyond 24 hours in patients with mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension (grade 1-2)

Exclusion Criteria:

* Severe hypertension
* Secondary hypertension
* Grade III/IV hypertensive retinopathy
* Type 1 diabetes
* Cerebrovascular or cardiovascular event during the last 12 months prior to inclusion.
* Pregnant or lactating females
* History of malignancy.
* shift workers
* intolerant to ABPM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy of valsartan by testing the hypothesis of superior 24 hrs diastolic BP lowering after missing dose compared with enalapril. | 16 weeks

SECONDARY OUTCOMES:
To demonstrate that valsartan is more effective than enalapril in terms of systolic 24 hrs BP lowering after missing dose. | 16 weeks
To show that valsartan is more effective than enalapril in reducing systolic and diastolic BP in the time interval 20-24 hours after dose administration. | 16 weeks
To show that valsartan has a more favorable effect than enalapril in smoothness index and through/peak ratio. | 16 weeks
To demonstrate that valsartan offers better safety profile than enalapril. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ramon C Hermida, Ph.D., Principal Investigator — University of Vigo
Locations (1):
- Hospital Clínico Universitario de Santiago, Santiago de Compostela, Spain

REFERENCES:
- [Derived] Hermida RC, Ayala DE, Khder Y, Calvo C. Ambulatory blood pressure-lowering effects of valsartan and enalapril after a missed dose in previously untreated patients with hypertension: a prospective, randomized, open-label, blinded end-point trial. Clin Ther. 2008 Jan;30(1):108-20. doi: 10.1016/j.clinthera.2008.01.012. PMID 18343247